CLINICAL TRIAL: NCT04695769
Title: The Role of Combined Ribavirin and Sofosbuvir/Velpatasvir/Voxilaprevir in Treatment of Chronic Hepatitis C Non-responders; A Randomized Controlled Trial
Brief Title: Combined Ribavirin With Sofosbuvir/Velpatasvir/Voxilaprevir in Retreatment of Chronic Hepatitis C Non-responders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mohammed Emadeldeen, Hepato-gastroenterology specialist, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HelwanU 76-2020
Record Dates: First submitted 2020-12-24; First posted 2021-01-05 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Chronic Hepatitis C
Keywords: HCV; Relapse; treatment failure
MeSH Terms: conditions — Hepatitis C, Chronic; Recurrence | interventions — Sofosbuvir; velpatasvir; voxilaprevir; sofosbuvir velpatasvir voxilaprevir drug combination; Ribavirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: SOF/VEL/VOX with RBV (Experimental): Drug: Sofosbuvir/Velpatasvir/Voxilaprevir 400/100/100 mg tablets (single pill combination administered orally once daily) plus Ribavirin (weight-based dose 1000 or 1200 mg daily according to patient body weight: < or > 60 kg).
  Another name: Vosevi, RBV
  Interventions: Drug: Sofosbuvir / Velpatasvir / Voxilaprevir Oral Tablet [Vosevi] plus Ribavirin
- Group B: SOF/VEL/VOX (Active Comparator): Drug: Sofosbuvir/Velpatasvir/Voxilaprevir 400/100/100 mg tablets (single pill combination administered orally once daily).
  Another name: Vosevi
  Interventions: Drug: Sofosbuvir / Velpatasvir / Voxilaprevir Oral Tablet [Vosevi]

INTERVENTIONS:
Drug: Sofosbuvir / Velpatasvir / Voxilaprevir Oral Tablet [Vosevi] plus Ribavirin — Patients will receive Sofosbuvir / Velpatasvir / Voxilaprevir with weight-based Ribavirin for 12 weeks.
  Other Names: Vosevi + RBV
  Arms: Group A: SOF/VEL/VOX with RBV
Drug: Sofosbuvir / Velpatasvir / Voxilaprevir Oral Tablet [Vosevi] — Patients will receive Sofosbuvir / Velpatasvir / Voxilaprevir for 12 weeks.
  Other Names: Vosevi
  Arms: Group B: SOF/VEL/VOX

SUMMARY:
This study aims to assess the role of ribavirin as an adjuvant to sofosbuvir/velpatasvir/voxilaprevir combination in retreatment of chronic hepatitis C with previous treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) patients with chronic hepatitis C and detectable HCV RNA by Polymerase Chain Reaction (PCR) after completion of previous direct-acting antiviral regimen, and eligible for antiviral treatment.

Exclusion Criteria:

* Patients with decompensated cirrhosis (Child-Pugh score B and C).
* Patients with platelet count less than 50000/ mm³.
* Patients with HCC or extrahepatic malignancy.
* Pregnancy or inability to use an effective contraceptive method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Achievement of sustained virological response (SVR) | 12 weeks post treatment
  Percentage of patients with Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12) SVR12 is defined as HCV RNA < the lower limit of quantitation 12 weeks following the last dose of study drug.

SECONDARY OUTCOMES:
Tolerability | During 12 weeks of treatment
  Tolerability assessment by reporting any adverse events in addition to laboratory abnormalities via continuous monitoring of CBC, transaminases, serum bilirubin, and serum creatinine at baseline and every 4 weeks during treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Helwan University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Kassas M, Emadeldeen M, Hassany M, Esmat G, Gomaa AA, El-Raey F, Congly SE, Liu H, Lee SS. A randomized-controlled trial of SOF/VEL/VOX with or without ribavirin for retreatment of chronic hepatitis C. J Hepatol. 2023 Aug;79(2):314-320. doi: 10.1016/j.jhep.2023.04.011. Epub 2023 Apr 23. PMID 37088312